CLINICAL TRIAL: NCT06533410
Title: Using the Chinese Indigenization FS Scale in the Diagnosis of Fibromyalgia： Specificity and Sensitivity in Clinical Practice
Status: Recruiting | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government); BAODING NO.1 HOSPITAL OF TCM (Unknown); Inner Mongolia Hospital of Traditional Chinese Medicine (Unknown); Shenzhen Hospital of Traditional Chinese Medicine (Unknown); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Juan Jiao, professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2024-121-KY
Record Dates: First submitted 2024-07-08; First posted 2024-08-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic widespread pain
  Interventions: Diagnostic Test: The FM Diagnosis and Assessment Scale will be filled out, and there will be no other interventions beyond that
- Fibromyalgia
  Interventions: Diagnostic Test: The FM Diagnosis and Assessment Scale will be filled out, and there will be no other interventions beyond that

INTERVENTIONS:
Diagnostic Test: The FM Diagnosis and Assessment Scale will be filled out, and there will be no other interventions beyond that — The FM Diagnosis and Assessment Scale will be filled out, and there will be no other interventions beyond that

SUMMARY:
This study aimed to evaluate the specificity and sensitivity of the diagnostic criteria for fibromyalgia after conducting local validation in China.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age; Patients with chronic widespread pain; Able to complete the questionnaire.

Exclusion Criteria:

* Terminal patients with severe psychiatric diseases, tumors, systemic lupus erythematosus, systemic sclerosis, or other serious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic widespread pain: pain on the left side of the body, pain on the right side, pain above the waist, and pain below the waist. In addition, axial bone pain (cervical or anterior chest or thoracic or lower back pain) must be present. In this definition, shoulder and hip pain are considered pain on each affected side. "Lower back pain" is thought to be lower pain.)
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of fibromyalgia with the Polysymptomatic Distress Scale(PDS) | up to 1 week
  The PDS scale fibromyalgia severity (FS) scale also known as the fibromyalgia severity (FS) scale. It is the sum of the WPI and SSS, and ranges is from 0-31 with higher score indicating more severity.

SECONDARY OUTCOMES:
QOL as measured by Short Form-36 Health Status Questionnaire(SF-36) | up to 1 week
  The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status
Fibromyalgia symptoms severity as measured by the Rebised Fibromyalgia Impact Questionnaire(FIQR) | up to 1 week
  The FIQR has 21 individual questions and is divided into three linked sets of domains as the FIQ (that is, function, overall impact and symptoms). It differs from the FIQ in having modified function questions and the inclusion of questions on memory, tenderness, balance and environmental sensitivity. The total FIQR is the sum of the three modified domain scores which ranges is also from 0-100 with higher score indicating more sever symptoms.
Depression scores as measured by Beck depression inventory(BDI) | up to 1 week
  The Beck II Depression Inventory (BDI) assesses the severity of depressive symptoms. Scores range from 0 to 39, with higher scores indicate a greater degree of depression severity.
Stress scores as measured by Perceived Stress Scale(PSS) | up to 1 week
  The Perceived Stress Scale (PSS) is for measuring the perception of stress and The Perceived Stress Scale (PSS) is for measuring the perception of stress and current levels of experienced stress. Scores range from 0 to 56, with higher total score indicating a greater degree of symptom severity
Sleep scores as measured by Pittsburgh sleep quality index(PSQI) | up to 1 week
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.
Fatigue was measured by the Multidimensional Fatigue Inventory(MFI-20) | up to 1 week
  The Multidimensional Fatigue Inventory-20 (MFI-20) measures fatigue severity. The MFI-20 total score ranges from 0 to 80, with higher scores indicate more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No